CLINICAL TRIAL: NCT06653010
Title: A Clinical Study on the Safety and Efficacy of Universal CAR-T Cells (REVO-UWD-01) for Metastatic Colorectal Cancer
Brief Title: Universal CAR-T Cells (REVO-UWD-01) for Metastatic Colorectal Cancer
Acronym: Wondercel-UWD1
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wondercel Biotech (ShenZhen) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-REVO-UWD-01
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: CRC (Colorectal Cancer); Metastatic Colorectal Cancer
Keywords: Universal CAR-T cells; Allogeneic CAR-T therapy; Wondercel REVO U-CAR platform; REVO-UWD-01
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose injection of REVO-UWD-01 (Experimental): Dose escalation will be performed for the single dose injection of REVO-UWD-01 for treating mCRC
  Interventions: Biological: Universal CAR-T cells injection for treating mCRC

INTERVENTIONS:
Biological: Universal CAR-T cells injection for treating mCRC — A novel universal CAR-T platform to treat cancer patients
  Other Names: Allogeneic CAR-T cells (REVO-UWD-01)

SUMMARY:
This is an investigator initiated trial to assess the efficacy and safety of a GCC-targeting CAR-T therapy (REVO-UWD-01) in the metastatic colorectal cancer. It also aims to explore the feasibility of using a novel universal CAR-T cell platform.

DETAILED DESCRIPTION:
The study will use T cells from healthy donors, modified using a novel universal CAR-T technology, to treat metastatic colorectal cancer patients. The antigen-binding site of the CAR molecule recognizes GCC as the target.

The main questions it aims to answer are:

* What is the maximum tolerated dose (MTD) of GCC-CAR-T therapy in universal CAR-T cell treatments?
* What are the dose-limiting toxicities (DLT) and treatment-emergent adverse events (TEAE)?
* What is the treatment's efficacy, as measured by objective response rate (ORR) and progression-free survival (PFS)? Researchers will assess whether universal CAR-T cells have good safety and efficacy in treating colorectal cancer, while improving accessibility and lowering treatment costs.

Participants will:

* Receive universal GCC-CAR-T cells through a 3+3 dose escalation scheme.
* Undergo chemotherapy conditioning before CAR-T infusion.
* Be monitored for adverse events, immune response, and disease progression.

The study will collect data on both short-term outcomes (within the first few months post-treatment) and long-term safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years and ≤75 years old.
2. Pathological Diagnosis: Pathologically confirmed metastatic colorectal cancer with radiographically confirmed metastatic lesions (e.g., CT or MRI).
3. GCC Expression: Tumor lesions assessed by immunohistochemistry (IHC) showing GCC expression ≥1+ in ≥50% of the area (randomly select at least 5 fields from tumor regions for evaluation; at least 5 unstained slides must be provided for assessment).
4. Measurable Lesions: At least one measurable lesion per RECIST 1.1 criteria; measurable lesions should not have received prior radiotherapy or interventional local therapy (lesions in previously irradiated or locally treated fields may be selected as target lesions if confirmed to have progressed).
5. Prior Treatment: Participants with advanced colorectal cancer who have progressed or are intolerant after ≥2 lines of standard therapy (with clear documentation).
6. ECOG Performance Status: 0 or 1.
7. Expected Survival: ≥90 days (as assessed by the investigator based on the participant's clinical condition).
8. Organ Function:
9. Absolute neutrophil count ≥1.5 × 10⁹/L;
10. Platelet count ≥80 × 10⁹/L;
11. Hemoglobin ≥9 g/dL;
12. Liver function:

    1. Total bilirubin ≤1.5 × ULN (≤2.0 × ULN for Gilbert's syndrome);
    2. AST and ALT ≤5 × ULN;
13. INR <1.3 (INR <3 for participants on anticoagulant therapy);
14. Serum creatinine ≤1.5 mg/dL (132.6 μmol/L) or eGFR ≥50 mL/min/1.73 m²;
15. Cardiac ejection fraction >50%.
16. Bleeding Risk: No active bleeding or bleeding tendency.
17. Fertility Requirements:
18. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment and agree to use effective contraception during treatment and for 8 weeks after the last dose;
19. Male participants must also use effective contraception during treatment and for 8 weeks after the last dose.
20. Informed Consent: Participants voluntarily enroll in the study, provide signed informed consent, demonstrate good compliance, and cooperate with follow-up.

Exclusion Criteria：

1. • Pregnant or breastfeeding women;
2. • Received chemotherapy, targeted therapy, monoclonal antibody therapy, or traditional Chinese medicine anti-tumor therapy within 14 days prior to cell collection;
3. • Participated in another drug clinical trial within 4 weeks prior to study initiation;
4. • Any of the following cardiovascular or cerebrovascular diseases or risk factors:
5. LVEF <50%;
6. NYHA Class III or IV heart failure;
7. History of myocarditis, cardiomyopathy, or myocardial infarction within 6 months prior to enrollment (unless cardiac function has recovered as confirmed by the investigator);
8. Uncontrolled arrhythmias (e.g., atrial fibrillation, ventricular tachycardia) or requiring long-term anti-arrhythmic therapy;
9. QTcF >480 ms on screening ECG;
10. Uncontrolled hypertension (systolic BP >160 mmHg or diastolic BP >100 mmHg);
11. History of ischemic or hemorrhagic stroke (unless stable for >6 months with no sequelae);
12. Uncontrolled intracranial lesions (e.g., brain tumors, aneurysms);
13. History of DVT or PE (unless on stable anticoagulant therapy for ≥6 months);
14. Significantly elevated troponin or BNP/NT-proBNP levels suggestive of potential cardiac injury or dysfunction;
15. • Non-healing wounds or fractures for a prolonged period;
16. • Coagulation disorders or bleeding diathesis;
17. • History of substance abuse (including psychiatric drugs) that cannot be discontinued or history of psychiatric disorders;
18. • Uncontrolled or active fungal, bacterial, viral, or other infections.
19. • Prior anti-tumor treatment-related toxicities not recovered to ≤Grade 1 or to levels specified in the inclusion/exclusion criteria;
20. • Known HIV infection; known active syphilis; or active hepatitis B (HBsAg-positive and HBV-DNA ≥500 IU/mL or above the lower limit of detection, whichever is higher) or hepatitis C (anti-HCV-positive and HCV-RNA above the lower limit of detection);
21. • Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage despite appropriate intervention;
22. • Severe allergic reaction history to key study treatments (including fludarabine, cyclophosphamide, mycophenolate sodium, tocilizumab, and anti-infective agents used during preconditioning);
23. • Active autoimmune disease requiring systemic treatment within 2 years (including but not limited to autoimmune hepatitis, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism); physiologic corticosteroid replacement therapy (e.g., thyroxine, insulin, or corticosteroids for adrenal or pituitary insufficiency) is not considered systemic treatment;
24. • Female participants unwilling to use contraception from informed consent through 6 months after CAR-T cell infusion;
25. • Participants with leptomeningeal metastasis, brainstem metastasis, spinal cord metastasis and/or compression, or active/symptomatic CNS metastases not treated locally;
26. • History of interstitial lung disease (ILD) or non-infectious pneumonitis requiring steroid treatment;
27. • Clinically significant pulmonary impairment due to lung comorbidities, including but not limited to underlying pulmonary disease (e.g., pulmonary embolism, severe asthma, or severe COPD within 3 months prior to enrollment), any autoimmune, connective tissue, or inflammatory disorders involving the lungs (e.g., rheumatoid arthritis, sarcoidosis), or prior pneumonectomy;
28. • Any condition deemed by the investigator to interfere with drug evaluation, participant safety, or study outcomes, or any other condition making the participant unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2027-10-20 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Within the first month post-infusion.
  The highest dose of GCC-CAR-T cells that can be administered without causing unacceptable side effects, measured during the dose escalation phase.
Dose-Limiting Toxicities (DLT) | Within the first month post-infusion.
  The incidence of treatment-related toxicities that prevent further dose escalation.
Treatment-Emergent Adverse Events (TEAE) | From the administration of UWD-01 CAR-T cells through six months post-infusion
  The frequency and severity of adverse events that arise following the administration of UWD-01-CAR-T cells.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Measured at 3 and 6 months after treatment.
  The proportion of patients with a measurable reduction in tumor size (complete or partial response) following GCC-CAR-T therapy.
Progression-Free Survival (PFS) | From the start of treatment up to 5 years.
  The length of time during and after treatment that the patient lives without disease progression.
Overall Survival (OS) | From the start of treatment up to maximum follow-up period of five years.
  The duration from the start of treatment to the time of death from any cause.
Duration of Response (DOR) | From the administration of UWD-01 CAR-T cells to a maximum follow-up period of five years.
  The time from initial tumor response (CR or PR) to disease progression or relapse or any cause of death.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shenzhen Nanshan People's Hospital, Shenzhen, Guangdong
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No